CLINICAL TRIAL: NCT06799312
Title: Comparative Effectiveness of Ipsilesional High-frequency rTMS, Contralesional Continuous Burst Theta rTMS, and Sham rTMS, Each Combined With Physiotherapy, in Subacute Ischemic Stroke Upper Limb Recovery : Clinical, Neurophysiological and Radiological: A Double-blinded Randomized Clinical Trial
Brief Title: Comparative Effectiveness of Ipsilesional High-frequency rTMS, Contralesional Continuous Burst Theta rTMS, and Sham rTMS, Each Combined With Physiotherapy, in Subacute Ischemic Stroke Upper Limb Recovery : Clinical, Neurophysiological and Radiological
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammad Ahmad Mohammad Korayem, Assisstant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NeuroRehabStroke2025
Record Dates: First submitted 2025-01-15; First posted 2025-01-29 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Repetitive Transcranial Magnetic Stimulation; Stroke; Functional MRI
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: A double blinded randomized controlled trial comparing different interventions on separate groups simultaneously.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both participants and investigators are blinded to the intervention type, with sham rTMS serving as the control for maintaining blinding integrity.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ipsilesional high frequency rTMS combined with physiotherapy (Active Comparator): rTMS Protocol:
  Stimulation delivered to the hand area of the ipsilesional primary motor cortex (M1).
  Frequency: 3 Hz.
  Stimulation: 2 seconds per train, 37 trains per session.
  Total pulses: 750 per session at 130% of the resting motor threshold (RMT).
  Physiotherapy:
  Patients receive standard physiotherapy sessions.
  Interventions: Device: Ipsilesional high frequency rTMS combined with physiotherapy
- Contralesional Continuous Burst Theta rTMS (cTBS) + Physiotherapy (Active Comparator): rTMS Protocol:
  Stimulation delivered to the contralesional primary motor cortex (M1).
  Protocol: Continuous bursts of 3 stimuli at 50 Hz, repeated at 5 bursts per second.
  Duration: 40 seconds per session.
  Stimulation intensity: 70% of RMT with a biphasic TMS-induced current at a 45° angle to the midline.
  Physiotherapy:
  Patients receive standard physiotherapy sessions.
  Interventions: Device: Contralesional Continuous Burst Theta rTMS (cTBS) + Physiotherapy
- Sham rTMS + Physiotherapy (Sham Comparator): Patients receive a sham stimulation designed to mimic rTMS without delivering active magnetic pulses.
  This maintains blinding for participants and investigators.
  Physiotherapy:
  Patients receive standard physiotherapy sessions.
  Interventions: Device: Sham rTMS + Physiotherapy

INTERVENTIONS:
Device: Ipsilesional high frequency rTMS combined with physiotherapy — As mentioned in details in arms description.
  Arms: Ipsilesional high frequency rTMS combined with physiotherapy
Device: Contralesional Continuous Burst Theta rTMS (cTBS) + Physiotherapy — As mentioned in details in arms description.
  Arms: Contralesional Continuous Burst Theta rTMS (cTBS) + Physiotherapy
Device: Sham rTMS + Physiotherapy — As mentioned in details in arms description.
  Arms: Sham rTMS + Physiotherapy

SUMMARY:
To compare the efficacy of lesional high-frequency rTMS, contralesional cTBS, and sham stimulation in improving motor and cognitive recovery in post-stroke patients undergoing physiotherapy.

DETAILED DESCRIPTION:
Globally, stroke is the second leading cause of both death and disability. In 2020, the global prevalence of all stroke subtypes was 89.13 million cases, with acute ischemic stroke (AIS) comprising 76.47% of these, equating to 68.16 million cases . AIS presents a major global public health concern, given the wide range of disabilities it causes, including cognitive impairments. Survivors of stroke bear a significant burden due to the persistent disability they experience over time . Immediately following a stroke, motor impairments are accompanied by significant alterations in the affected primary motor cortex (M1) - detected by transcranial magnetic stimulation (TMS)- resulting in reduced cortical excitability. This can be evidenced by the absence of recordable motor evoked potentials (MEPs), diminished MEP amplitudes, and increased resting motor threshold (rMT). Additionally, stroke can alter brain connectivity, particularly in terms of functional connectivity, which has implications for recovery. Neuroplasticity plays a crucial role in recovery after stroke, allowing the brain to reorganize and compensate for lost functions. Physiotherapy is a cornerstone of post-stroke rehabilitation, particularly for upper limb recovery and cognitive improvement, with early intervention associated with better outcomes. Repetitive transcranial magnetic stimulation (rTMS) has shown promise in the early stages post-stroke, enhancing motor and cognitive recovery, particularly when applied within two weeks of stroke onset. MEPs can be used to monitor changes in cortical excitability and have been linked to both cognitive and motor recovery. Combining rTMS with diffusion tensor imaging (DTI) allows for the assessment of both functional and structural brain changes, providing a deeper understanding of rTMS's therapeutic effects. DTI, through fractional anisotropy (FA), helps to evaluate white matter integrity, and studies have shown that increased FA correlates with motor recovery, making it a valuable tool in examining the structural changes induced by rTMS in stroke recovery. While high frequency rTMS targeting the ipsilesional motor cortex (M1) has demonstrated efficacy in enhancing motor recovery, contralesional continuous theta-burst stimulation (cTBS) has shown promising results offering an alternative by modulating interhemispheric inhibition. However, no studies have directly compared the efficacy of these two paradigms against each other and sham stimulation in subacute stroke recovery. This study seeks to address this gap by comparing the outcomes of lesional high frequency rTMS, contralesional cTBS, and sham stimulation in combination with physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* First-ever ischemic stroke, confirmed by imaging.
* Stroke affecting the non-dominant hemisphere (cortical or subcortical) within the middle cerebral artery (MCA) territory.
* Acute to subacute stage of stroke (time since onset: 48 hours to 2 weeks).
* Ability to comply with the study protocol and interventions.

Exclusion Criteria:

* Hemorrhagic stroke or bilateral stroke.
* Severe cognitive impairment, defined as a Montreal Cognitive Assessment (MoCA) score < 10.
* Contraindications to TMS, such as: History of epilepsy, Metallic implants in the head, Other contraindications based on TMS safety guidelines.
* Comorbid conditions that limit participation in rehabilitation.
* Severe neglect or aphasia that would impede participation in therapy.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Score in Nottingham Sensory Assessment in points | Within the time frame of the study , around 18 months
Score in modified Ashworth Scale in points | Within the time frame of the study , around 18 months
Score in Fugl-Meyer assessment scale in points | Within the time frame of the study , around 18 months

SECONDARY OUTCOMES:
Cortical Excitability Improvement | Within the time frame of the study , around 18 months
  Evaluates changes in cortical excitability parameters (e.g., resting motor threshold measured in Percentage of maximum stimulator output , cortical silent period measured in milliseconds, transcallosal inhibition measured in milliseconds) using TMS after intervention.
Enhancement of White Matter Integrity | Within the time frame of the study , around 18 months
  Assesses changes in white matter integrity using functional MRI.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://dx.doi.org/10.1016/S1474-4422(19)30034-1
- See also: Related Info — http://dx.doi.org/10.4103/0972-2327.168631
- See also: Related Info — http://dx.doi.org/10.1016/j.brs.2017.03.008
- See also: Related Info — http://dx.doi.org/10.1016/j.nicl.2020.102538
- See also: Related Info — https://www.ncbi.nlm.nih.gov/books/NBK551707/
- See also: Related Info — http://dx.doi.org/10.21037/apm-21-3710
- See also: Related Info — http://dx.doi.org/10.1186/s12883-024-03565-8
- See also: Related Info — http://dx.doi.org/10.1016/j.nrl.2016.03.008
- See also: Related Info — http://dx.doi.org/10.3389/fneur.2019.01269
- See also: Related Info — https://doi.org/10.3389/fnbeh.2018.00160
- See also: Related Info — https://doi.org/10.1016/j.clinph.2009.08.016
- See also: Related Info — https://doi.org/10.15453/2168-6408.1164